CLINICAL TRIAL: NCT05905406
Title: Effect of Femoral Quadriceps Muscle Length on Fatigue, Neuromuscular Performance, Oxygen Uptake and Discomfort Induced by Neuromuscular Electrical Stimulation
Brief Title: Effect of Femoral Quadriceps Muscle Length on Fatigue Induced by Neuromuscular Electrical Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Physical Therapist Assistant Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68446223.2.0000.80
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Electrical Stimulation
Keywords: Electrical Stimulation; Fatigue; Electromyographic activity; Muscular architecture; Tendinous properties; Extraction of oxygen
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- S60 (Experimental): The Hip will be positioned at 80°, and knee positioned 60°. The sessions will be initiated with heating and muscle enhancement. The following outcomes will be observed before and after the fatigue protocol: (1) CVIM; (2) voluntary activation level; (3) electromyographic activity; (4) muscular architecture; and (5) tendinous properties. During the fatigue protocol, except for item 1), will be evaluated: (1) fatigue by torque decay curve; (2) integral force-time; (3) muscular architecture; (4) tendinous properties; and tissue oxygen extraction.
  Interventions: Other: Electrical estimulation
- S20 (Experimental): The Hip will be positioned at 80°, and knee positioned 20°. The sessions will be initiated with heating and muscle enhancement. The following outcomes will be observed before and after the fatigue protocol: (1) CVIM; (2) voluntary activation level; (3) electromyographic activity; (4) muscular architecture; and (5) tendinous properties. During the fatigue protocol, except for item 1), will be evaluated: (1) fatigue by torque decay curve; (2) integral force-time; (3) muscular architecture; (4) tendinous properties; and tissue oxygen extraction.
  Interventions: Other: Electrical estimulation
- D60 (Experimental): The Hip will be positioned at 0°, and knee positioned 60°. The sessions will be initiated with heating and muscle enhancement. The following outcomes will be observed before and after the fatigue protocol: (1) CVIM; (2) voluntary activation level; (3) electromyographic activity; (4) muscular architecture; and (5) tendinous properties. During the fatigue protocol, except for item 1), will be evaluated: (1) fatigue by torque decay curve; (2) integral force-time; (3) muscular architecture; (4) tendinous properties; and tissue oxygen extraction.
  Interventions: Other: Electrical estimulation
- D20 (Experimental): The Hip will be positioned at 0°, and knee positioned 20°. The sessions will be initiated with heating and muscle enhancement. The following outcomes will be observed before and after the fatigue protocol: (1) CVIM; (2) voluntary activation level; (3) electromyographic activity; (4) muscular architecture; and (5) tendinous properties. During the fatigue protocol, except for item 1), will be evaluated: (1) fatigue by torque decay curve; (2) integral force-time; (3) muscular architecture; (4) tendinous properties; and tissue oxygen extraction.
  Interventions: Other: Electrical estimulation

INTERVENTIONS:
Other: Electrical estimulation — Electrical estimulation during the fatigue protocol. Frequency = 100 Hz, pulse duration = 500 µs, time ON = 20 s (including rise time = 1.0 s and descent time = 1.0 s) and off time = 20 sec

SUMMARY:
This study aims To investigate the effects of Quadriceps femoris muscle length on neuromuscular fatigue induced by NMES, muscle performance, discomfort and peripheral oxygen extraction.

DETAILED DESCRIPTION:
This is a crossover, experimental, randomized and double-blind trial (participant and statistician). The procedures will be performed at the Neuromuscular Performance Laboratory and the Musculotendineal Plasticity Laboratory (LaPlasT) of the Faculty of Ceilândia/University of Brasília to evaluate the neuromuscular fatigue generated during NMES of the QF muscle in different muscle lengths, according to the articular angles of the hip and knee. Participants aged between 18 and 45 years of age, of both sexes, healthy, with body mass index (BMI) between 18.5 and 24.9 kg/ m² (ie eutrophic), who did not perform systematic training to strengthen the lower limbs in the last six months, practitioners or not of recreational sports activities, physically active according to the International Physical Activity Questionnaire (IPAQ), and with minimum torque reach of 20% of MVC during NMES without excessive discomfort. Those who have: edema, dermal injury, limitation of the range of joint motion, deformity or amputation in any part of the lower limbs, as well as a history of patellar dislocation or trauma to the lower limbs or trunk that compromises the results. Also excluded are those with conditions that affect musculotendineal morphology or neuromuscular excitability such as diabetes mellitus type II, familial hypercholesterolemia, neuromuscular disease and severe cardiopathy, or conditions that procedures, such as cognitive impairment, psychiatric disease, chemical dependence or behavioral problems (Dudley-Javoroski et al., 2010). Participants will be initially familiar with assessments and training with EENM. In familiarization, will be performed: Antropometry (height and body mass); location of the motor points; randomization of the order of articular positioning that will be evaluated; muscle enhancement; and three CVIM. The fatigue protocol with NMES will occur at 20% of MVC in positions: bench press with knee at 60º of flexion (Sup60), sitting with knee at 60º (Sen60), bench press at 20º (Sup20) and Sitting with knee at 20º (Sen20). These positions were chosen considering that: (1) SJ60 is the position in which the knee angle provides the optimal QF length for maximum torque production (Scott et al., 2019), and the hip angle provides a neutral length for the RF (Bampouras et al., 2017); (2) QF is commonly stimulated with knees fully extended (Fitzgerald et al., 2003). However, with the knees extended, it is not possible to measure the extensor torque of the knee properly in the isokinetic dynamometer (Babault et al., 2003). Therefore, we chose 20º knee flexion as an approximate position; (3) the hip angle affects the length of RF and myotendinous stiffness of QF (Bampouras et al., 2017), so the knee angles (60º and 20º) will be evaluated with the participants both seated (hip in flexion; 85º) when lying down (hip in extension; 0º). During familiarization, for anthropometric assessment (height, body mass and BMI), participants will be barefoot and wearing light clothes. The BMI will be obtained by the ratio of the weight of the participants in kilos with the square of the height (kg/m2). To determine the level of engagement in physical activities, the IPAQ will be applied, which contains 7 items that assess the frequency (days) and duration (minutes and/ or hours) spent on physical activities in the last week (Scholes et al., 2016). After familiarization, there will be four sessions of fatigue induced by NMES, composed of 20 electrically induced contractions at 20% of CVM (CEI20%). Each session will be as confirmed by the volunteer regarding the absence of any residual muscle discomfort arising from the previous session. The sessions will be initiated with heating and muscle enhancement. The following outcomes will be observed before, during and after the fatigue protocol: CVIM; reflex H, Wave M and voluntary activation level; electromyographic activity; muscular architecture; tendinous properties and tissue oxygen extraction. During the fatigue protocol (five first and five last evoked contractions, will be evaluated: (1) fatigability by the torque decay curve; (2) integral force-time; (3) tissue extraction of oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 45 years of age;
* Both sexes;
* Healthy;
* Body mass index (BMI) between 18.5 and 24.9 kg/ m² (ie eutrophic);
* Who did not perform systematic training strengthening of the lower limbs in the last six months;
* Practitioners or not of recreational sports activities;
* Physically active according to the International Physical Activity Questionnaire (IPAQ);
* Who with minimum torque reach of 20% of MVC during NMES without excessive discomfort.

Exclusion Criteria:

* Edema;
* Dermal injury;
* Limitation of the range of joint motion;
* Deformity or amputation in any part of the lower limbs, as well as a history of patellar dislocation or trauma to the lower limbs or trunk that compromises the results;
* Those with conditions that affect musculotendineal morphology or neuromuscular excitability such as diabetes mellitus type II, familial hypercholesterolemia, neuromuscular disease and severe cardiopathy;
* Conditions that make it impossible to cooperate with procedures, such as cognitive impairment, psychiatric illness, chemical dependence or behavioral problems.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | an average of 1 year and half
  Fatigue index evoked by electrical stimulation

SECONDARY OUTCOMES:
Reflex H | an average of 1 year and half
  Analysis of the physiologic variables
M wave | an average of 1 year and half
  Analysis of the physiologic variables
Voluntary activation level | an average of 1 year and half
  Analysis of the physiologic variables
Surface electromyographic activity (EMG) | an average of 1 year and half
  Level of activation of muscle
Muscle thickness | an average of 1 year and half
  Datas from Muscle architecture
Displacement of the tendon-aponeurosis complex | an average of 1 year and half
  Datas from Muscle architecture
Muscle stiffness | an average of 1 year and half
  Datas from Muscle architecture
Properties of the patellar tendon | an average of 1 year and half
  cross section area from patellar tendon
Oxidized hemoglobin (Oxy-[Hb/Mb]) | an average of 1 year and half
  tissue extraction
Deoxidized hemoglobin (deoxy-[Hb/Mb]) | an average of 1 year and half
  tissue extraction
Total hemoglobin (total-[Hb/Mb]) | an average of 1 year and half
  tissue extraction
Sensorial discomfort during all phases in protocol | an average of 1 year and half
  Sensorial discomfort assessed by VAS

IPD SHARING:
Plan to Share IPD: No
The authors consider sharing the data depending on the situation

REFERENCES:
- [Background] Ando R, Nosaka K, Inami T, Tomita A, Watanabe K, Blazevich AJ, Akima H. Difference in fascicle behaviors between superficial and deep quadriceps muscles during isometric contractions. Muscle Nerve. 2016 May;53(5):797-802. doi: 10.1002/mus.24905. Epub 2016 Mar 1. PMID 26355494
- [Background] Babault N, Cometti G, Bernardin M, Pousson M, Chatard JC. Effects of electromyostimulation training on muscle strength and power of elite rugby players. J Strength Cond Res. 2007 May;21(2):431-7. doi: 10.1519/R-19365.1. PMID 17530954
- [Background] Blazevich AJ. Effects of physical training and detraining, immobilisation, growth and aging on human fascicle geometry. Sports Med. 2006;36(12):1003-17. doi: 10.2165/00007256-200636120-00002. PMID 17123325
- [Background] Cavalcante JGT, de Almeida Ventura A, de Jesus Ferreira LG, de Sousa AMM, de Sousa Neto IV, de Cassia Marqueti R, Babault N, Durigan JLQ. Hip and Knee Joint Angles Determine Fatigue Onset during Quadriceps Neuromuscular Electrical Stimulation. Appl Bionics Biomech. 2022 Jul 22;2022:4612867. doi: 10.1155/2022/4612867. eCollection 2022. PMID 35937098
- [Background] Cavalcante JGT, Marqueti RC, Geremia JM, de Sousa Neto IV, Baroni BM, Silbernagel KG, Bottaro M, Babault N, Durigan JLQ. The Effect of Quadriceps Muscle Length on Maximum Neuromuscular Electrical Stimulation Evoked Contraction, Muscle Architecture, and Tendon-Aponeurosis Stiffness. Front Physiol. 2021 Mar 29;12:633589. doi: 10.3389/fphys.2021.633589. eCollection 2021. PMID 33854439
- [Background] Herzog W, Abrahamse SK, ter Keurs HE. Theoretical determination of force-length relations of intact human skeletal muscles using the cross-bridge model. Pflugers Arch. 1990 Apr;416(1-2):113-9. doi: 10.1007/BF00370231. PMID 2352828
- [Background] Kubo K, Ohgo K, Takeishi R, Yoshinaga K, Tsunoda N, Kanehisa H, Fukunaga T. Effects of isometric training at different knee angles on the muscle-tendon complex in vivo. Scand J Med Sci Sports. 2006 Jun;16(3):159-67. doi: 10.1111/j.1600-0838.2005.00450.x. PMID 16643193
- [Background] Maffiuletti NA. Physiological and methodological considerations for the use of neuromuscular electrical stimulation. Eur J Appl Physiol. 2010 Sep;110(2):223-34. doi: 10.1007/s00421-010-1502-y. Epub 2010 May 15. PMID 20473619
- [Background] Raiteri BJ. Aponeurosis behaviour during muscular contraction: A narrative review. Eur J Sport Sci. 2018 Sep;18(8):1128-1138. doi: 10.1080/17461391.2018.1472299. Epub 2018 May 28. PMID 29806988
- [Background] Talbot LA, Gaines JM, Ling SM, Metter EJ. A home-based protocol of electrical muscle stimulation for quadriceps muscle strength in older adults with osteoarthritis of the knee. J Rheumatol. 2003 Jul;30(7):1571-8. PMID 12858461